CLINICAL TRIAL: NCT02416518
Title: Genetic Exploration of the Molecular Basis of Malignancy in Adults
Acronym: GEMMA
Status: Completed | Type: Observational
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Other Study IDs: SH GEMMA
Record Dates: First submitted 2014-08-15; First posted 2015-04-15 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Neoplasms
Keywords: Cancer; Malignancy; Genomic; Molecular
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Genetic Exploration of the Molecular Basis of Malignancy in Adults.

DETAILED DESCRIPTION:
This protocol is not designed as a treatment protocol. Patients enrolled on this study will be treated according to the treating physician's plan of care, independent of enrollment into the study. Once enrolled, the physician may proceed with the appropriate plan of care during the period of specimen analysis if indicated. Upon return of the results, therapy may or may not be altered based upon the patient's pathology, pertinent medical and treatment history, imaging studies, available clinical trials, and on the CLIA validated clinical molecular profiling results. Regardless of the results, the patient will be offered a treatment selected on an empirical basis by the treating physician at the individual site. All patients enrolled in the study will be followed for clinical outcome. Clinical molecular profiling results will expire 14 weeks following the date the Foundation One report is received. No investigational agents will be administered as part of this study. However, patients may be referred to open clinical trials based on the results of profiling. Patients referred for clinical trial may receive investigational agents under a separate clinical trial in accordance with the written protocol for which they are subsequently enrolled. All anti-neoplastic drugs used while participating in this study, whether used on-label or off-label, will be administered to the patient by the route of administration published in the FDA approved package insert. In addition, the dosing of the agent (including dose modifications) will be calculated based upon what is published in the FDA approved package insert.

ELIGIBILITY:
Inclusion Criteria:

* Understand and provide written informed consent and HIPAA Authorization prior to initiation of any study-specific procedures.
* Have a life expectancy of >3 months.
* Have a diagnosis of metastatic, incurable cancer and have progressed on at least one line of systemic therapy OR a cancer with no standard 1st-line systemic therapy shown to prolong survival (or where a clinical trial recommended as the 1st-line option). Patients do not have to be off-treatment when enrolled on this trial. However, please see section 6.4.8 regarding the required wash-out period before starting any FDA approved on-label or off-label treatment.
* Measurable disease (RECIST 1.1).
* Be ≥18 years of age.
* ECOG Performance status 0 or 1.
* In the opinion of the investigator, be medically suitable for and willing to undergo a biopsy or surgical procedure to obtain tissue as a part of routine care for their malignancy OR have adequate archival tissue from a previous biopsy, performed no more than 14 weeks prior to enrollment, available for profiling.
* Have adequate organ and bone marrow function as defined below: Bone marrow: absolute neutrophil count (ANC) ≥ 1.5 x 109/L; hemoglobin ≥ 9 g/dL; platelets >100 x 109/L Renal: creatinine clearance ≥ 60 mL/min (calculated according to Cockcroft and Gault formula) or creatinine ≤ 1.5 mg/dL Hepatic: bilirubin ≤ 2.5 x the upper limit of normal (ULN); aspartate transaminases (AST/SGOT); alanine transaminases (ALT/SGPT) ≤ 2.5 x ULN (or ≤ 5 x ULN if due to underlying liver metastases)
* Female patients of childbearing potential must have a negative pregnancy test and agree to use at least two forms of contraception during the study and for at least one month after treatment discontinuation. For the purposes of this study, a female with child- bearing potential is defined as: any woman who meets the following criteria.

Has not undergone a hysterectomy or bilateral oophorectomy. Has not been naturally postmenopausal for at least 24 months (i.e. has had a menses at any time in the preceding 24 consecutive months).

* Male patients must use a form of barrier contraception that contains spermicide and is approved by the investigator / treating physician during the study and for at least one month after treatment discontinuation.
* No more than one prior screening attempt for SH GEMMA.

Exclusion Criteria:

* Have lesions that are not accessible to biopsy or not planned for biopsy as part of routine care OR if archival tissue will be used for profiling, an insufficient amount is available OR archival tissue was obtained ≥ 14 weeks prior to enrollment.
* Have diagnosis of a hematologic malignancy.
* Diagnosis of astrocytoma, glioblastoma multiforme, or any other primary brain cancer.
* Have concurrent uncontrolled malignancy.
* Have symptomatic CNS metastasis. Patients with a history of CNS metastases who have been treated with whole brain irradiation must be stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable dose of steroids for ≥ 2 weeks prior to enrollment.
* Have uncontrolled concurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent.
* Have known HIV, HBV, HCV infection.
* Previous enrollment in the SH GEMMA study. Patients are allowed one prior screening attempt.
* Are pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic, incurable cancer or cancer with no standard 1st-line systemic therapy that has shown prolonged survival
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-05; Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Feasibility (proportion of patients with successful molecular profiling compared to the number of patients enrolled) | 12 months
  Assess the feasibility of integrating genomic profiling in the adult oncology clinic within a community-based, multi-facility, health system. Feasibility is defined as the proportion of patients with successful molecular profiling compared to the number of patients enrolled.

SECONDARY OUTCOMES:
Patient and biopsy characteristics (including cancer type, biopsy type, and number of prior treatments) | 12 months
  Determine patient and biopsy characteristics, including cancer type, biopsy type, and number of prior treatments
Molecular testing characteristics (include: the frequency at which molecular analysis yields a genetic alteration, frequency of actionable alterations, and time from biopsy to final report) | 12 months
  Define molecular testing characteristics.This will include: the frequency at which molecular analysis yields a genetic alteration, frequency of actionable alterations, and time from biopsy to final report.
Molecular profiling influence | 12 months
  Determine how often molecular profiling influences treatment decision.Treatment type implemented will be classified as: standard therapy per treating physician, FDA approved off-label influenced by molecular profiling, internal targeted agent clinical trial influenced by molecular profiling, or external targeted agent clinical trial influenced by molecular profiling.
Clinical outcome of genomic based therapy (response according to RECIST 1.1 response criteria) | At 16wks following initiation of treatment impacted by molecular profiling. After 16wks tumor assessments per routine practice/clinical trial protocol requirements, continued until progression/time of treatment discontinuation, whichever is later.
  Determine the clinical outcome of genomic based therapy, as defined by response rate (according to RECIST 1.1 response criteria) the percent of patients with progression-free survival (PFS) at 4 months, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Powell, MD, Principal Investigator — Sanford Health; Anu Gaba, MD, Principal Investigator — Sanford Health; John Reynolds, MD, Principal Investigator — Sanford Health; Jayan Nair, MD, Principal Investigator — Sanford Health
Locations (4):
- United States (4):
  - Sanford Health, Bemidji, Minnesota
  - Sanford Health, Bismarck, North Dakota
  - Sanford Health, Fargo, North Dakota
  - Sanford Health, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No